CLINICAL TRIAL: NCT04940078
Title: Investigation of Pharmacokinetics Following Co-administration of Cagrilintide (NNC0174-0833) and Semaglutide Versus Separate Injections in Subjects With Overweight or Obesity
Brief Title: A Research Study to Compare Blood Levels of Cagrilintide and Semaglutide After Combined Versus Separate Injections in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-4614; U1111-1250-7789 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Intervention Model Description: The trial consists of a Part A with multiple weekly dosings at site and a Part B with a single dose (SD) part of the first dose step in Part A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: Cagrilintide and semaglutide in separate syringes (Experimental): Participants will up-titrated for 14 weeks (dose escalation every 4 weeks and 2 weeks at last dose escalation step prior to randomisation) with cagrilintide and semaglutide administered as separate injections. Followed by 8 weeks treatment with cagrilintide and semaglutide administered as separate injections. The 8-week treatment period covers 2 different doses of cagrilintide and semaglutide (1.7/1.7 mg and 2.4/2.4 mg with 4 weeks on each dose combination). Followed by a 38 days follow-up period.
  Interventions: Drug: Cagrilintide; Drug: semaglutide
- Part A: Cagrilintide and semaglutide combined in DV3384 device (Experimental): Participants will be up-titrated for 14 weeks (dose escalation every 4 weeks and 2 weeks at last dose escalation step prior to randomisation) with cagrilintide and semaglutide administered as separate injections. Followed by 8 weeks of treatment with cagrilintide and semaglutide administered using the DV3384 manual syringe. The 8-week treatment period covers 2 different doses of cagrilintide and semaglutide (1.7/1.7 mg and 2.4/2.4 mg with 4 weeks on each dose combination. Followed by a 38 days follow-up period.
  Interventions: Drug: Cagrilintide and semaglutide
- Part B: Cagrilintide and semaglutide combined in DV3384 device (Experimental): Participants will receive a single injection of Cagrilintide 0.25 mg/semaglutide 0.25 mg using the DV3384 manual syringe followed by a 28 days follow-up period.
  Interventions: Drug: Cagrilintide and semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Once weekly doses of cagrilintide gradually increased to 1.7 mg over 14 weeks and 2.4 mg s.c. for 2 weeks
  Arms: Part A: Cagrilintide and semaglutide in separate syringes
Drug: semaglutide — Once weekly doses of semaglutide gradually increased to 1.7 mg over 14 weeks and 2.4 mg s.c. over 2 weeks
  Arms: Part A: Cagrilintide and semaglutide in separate syringes
Drug: Cagrilintide and semaglutide — Cagrilintide and semaglutide combined and administered using the DV3384 manual syringe
  Arms: Part A: Cagrilintide and semaglutide combined in DV3384 device; Part B: Cagrilintide and semaglutide combined in DV3384 device

SUMMARY:
This study will compare two different ways of giving cagrilintide and semaglutide for treating overweight and obesity. The medicines will either be given together in 1 injection or as 2 separate injections.

The aim of the study is to find out how the different ways of injection affect the level of the medicines in the blood.

For the first 14 weeks of the study, participants will get cagrilintide and semaglutide as 2 separate injections. Then participants will either switch to getting the medicines as a combined injection or continue to get the separate injections for 8 weeks. Which treatment participants get after the first 14 weeks is decided by chance.

Participants will get the study medicines once a week for 22 weeks. A study nurse at the clinic will inject the medicines with a thin needle in participants stomach area.

The study will last for about 8 months.Participants will have 28 clinic visits with the study staff. For 4 of these visits, participants will stay in the clinic for 5 nights.

Participants will have blood drawn at 21 visits. Participants will have clinical assessments and participants will be asked about their health, medical history and habits including mental health questionnaires.

For women: Participants must not be able to become pregnant if they wish to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential (NCBP)
* Aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 27.0 and 39.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator

Exclusion Criteria:

* Previous participation in trial(s) with an amylin analogue unless documented that the subject was assigned to placebo treatment. Participation is defined as randomisation
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
AUC0-168h,cagri,2.4/2.4mg,SS area under the cagrilintide concentration-time curve during a dosing interval (0-168 hours) at steady state after last dosing of cagrilintide 2.4 mg in combination with semaglutide 2.4 mg | Day 148 (pre-dose) to Day 155 (168 hours post-dose)
  measured in nmol⸱h/L
Cmax,cagri,2.4/2.4mg,SS maximum concentration of cagrilintide at steady state after last dosing of cagrilintide 2.4 mg in combination with semaglutide 2.4 mg | Day 148 (pre-dose) to Day 155 (168 hours post-dose)
  measured in nmol/L
AUC0-168h,sema,2.4/2.4mg,SS area under the semaglutide concentration-time curve during a dosing interval (0-168 hours) at steady state after last dosing of semaglutide 2.4 mg in combination with cagrilintide 2.4 mg | Day 148 (pre-dose) to Day 155 (168 hours post-dose)
  measured in nmol⸱h/L
Cmax,sema,2.4/2.4mg,SS maximum concentration of semaglutide at steady state after last dosing of semaglutide 2.4 mg in combination with cagrilintide 2.4 mg | Day 148 (pre-dose) to Day 155 (168 hours post-dose)
  measured in nmol/L

SECONDARY OUTCOMES:
tmax,cagri,2.4/2.4mg,SS time since last dosing to maximum concentration of cagrilintide at steady state after last dosing of cagrilintide 2.4 mg in combination with semaglutide 2.4 mg | Day 148 (pre-dose) to Day 155 (168 hours post-dose)
  measured in hours
t½,cagri,2.4/2.4mg,SS terminal half-life of cagrilintide at steady state after last dosing of cagrilintide 2.4 mg in combination with semaglutide 2.4 mg | Day 148 (pre-dose) to Day 186 (912 hours post-dose)
  measured in hours
tmax,sema,2.4/2.4mg,SS time since last dosing to maximum concentration of semaglutide at steady state after last dosing of semaglutide 2.4 mg in combination with cagrilintide 2.4 mg | Day 148 (pre-dose) to Day 155 (168 hours post-dose)
  measured in hours
t½,sema,2.4/2.4mg,SS terminal half-life of semaglutide at steady state after last dosing of semaglutide 2.4 mg in combination with cagrilintide 2.4 mg | Day 148 (pre-dose) to Day 186 (912 hours post-dose)
  measured in hours
AUC0-168h,cagri,1.7/1.7mg,SS area under the cagrilintide concentration-time curve during a dosing interval (0-168 hours) at steady state after last dose of cagrilintide 1.7 mg in combination with semaglutide 1.7 mg | Day 120 (pre-dose) to Day 127 (168 hours post-dose)
  measured in nmol⸱h/L
AUC0-168h,sema,1.7/1.7mg,SS area under the semaglutide concentration-time curve during a dosing interval (0-168 hours) at steady state after last dose of semaglutide 1.7 mg in combination with cagrilintide 1.7 mg | Day 120 (pre-dose) to Day 127 (168 hours post-dose)
  measured in nmol⸱h/L
PART A: Number of treatment emergent adverse events | From time of dosing (Day 1) to follow-up (Day 186)
  count
PART B: Number of treatment emergent adverse events | From time of dosing (Day 1) to follow-up (Day 29)
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Altasciences Company Inc., Montreal, Quebec, Canada
- Novo Nordisk Investigational Site, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com